CLINICAL TRIAL: NCT00799812
Title: Test for Pre Operative Skin Preparations: ChloraPrep Triple Swabsticks, Hibiclens and Sterile Triple Swabsticks (Using Sterile Deionized Water)
Brief Title: Test for Pre Operative Skin Preparations
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: C. R. Bard (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: ENT 371-121
Record Dates: First submitted 2008-11-26; First posted 2008-12-01 (Estimated); Results first posted 2021-05-27 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-11

CONDITIONS: Topical Antisepsis
Keywords: antimicrobial; antisepsis
MeSH Terms: interventions — Chromogranins; chlorhexidine gluconate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- CHG Swabstick (3 @ once) (Experimental): Chlorhexidine gluconate (CHG) 2% w/v CHG/isopropyl alcohol (IPA) 70% v/v - 3 swabsticks applied @ same time
  Interventions: Drug: CHG 2% w/v & IPA 70% v/v, swabstick (3 @ once).
- CHG Swabstick sequential (Experimental): Chlorhexidine gluconate (CHG) 2% w/v and isopropyl alcohol (IPA) 70% v/v - 3 swabsticks applied sequentially
  Interventions: Drug: CHG 2% w/v & IPA 70% v/v swab applied sequentially
- Hibiclens (Active Comparator): Chlorhexidine gluconate (CHG) 4% w/v in an aqueous base
  Interventions: Drug: Aqueous CHG 4% w/v applied according to mfr's directions
- Sterile water swab (3 @ once) (Placebo Comparator): Sterile swabstick wetted with sterile deionized water - 3 swabsticks applied at the same time.
  Interventions: Other: Sterile swabstick with sterile water (3 @ once)
- Sterile water swabstick (sequential) (Placebo Comparator): Sterile swabstick wetted with sterile water--3 swabsticks applied sequentially.
  Interventions: Other: Sterile swabstick with sterile water (one-at-a-time)

INTERVENTIONS:
Drug: CHG 2% w/v & IPA 70% v/v, swabstick (3 @ once). — 3 swabsticks topically applied at the same time to intact skin
  Other Names: ChloraPrep Swabstick
  Arms: CHG Swabstick (3 @ once)
Drug: CHG 2% w/v & IPA 70% v/v swab applied sequentially — Chlorhexidine gluconate 2% w/v and isopropyl alcohol 70% v/v; 3 swabsticks applied sequentially to intact skin.
  Other Names: ChloraPrep Swabstick
  Arms: CHG Swabstick sequential
Drug: Aqueous CHG 4% w/v applied according to mfr's directions — Chlorhexidine gluconate 4% w/v in an aqueous base applied according to mfr's directions. Step 1) 5 ml of Hibiclens applied to a sterile gauze pad. Step 2) Product applied to treatment area on intact skin for 2 minutes. Area dried with sterile towel or sterile gauze. Steps 1 and 2 repeated.
  Other Names: Hibiclens
  Arms: Hibiclens
Other: Sterile swabstick with sterile water (3 @ once) — 3 sterile swabsticks wetted with sterile water topically applied to intact skin at the same time.
  Arms: Sterile water swab (3 @ once)
Other: Sterile swabstick with sterile water (one-at-a-time) — Sterile swabsticks wetted with sterile water topically applied to intact skin one-at-a-time.
  Arms: Sterile water swabstick (sequential)

SUMMARY:
Compare 2 application techniques of ChloraPrep Swabstick--3 swabsticks at once versus 3 swabsticks used sequentially. Hibiclens applied according to the manufacturer's directions. Sterile swabsticks (wetted with sterile deionizd water) applied using the same method as the ChloraPrep Swabstick.

DETAILED DESCRIPTION:
Determine differences (if any) in 2 different application techniques of ChloraPrep Swabstick--3 swabsticks at once versus 3 swabsticks used sequentially. Hibiclens, a liquid antibacterial soap, applied according to the manufacturer's directions as a active/positive comparison. Sterile swabsticks (wetted with sterile deionized water) applied as a negative comparison using the same method as the ChloraPrep swabstick.

Study uses topical sampling from the abdomen and the groin on intact skin and evaluates the germs left on the skin after treatment with ChloraPrep Swabsticks.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must read and sign an Informed Consent Form and be cooperative.
* Subjects must be in good general health.
* Subjects must have skin within 6 inches of the test site that is free of tattoos, dermatoses, abrasions, cuts, lesions, or other skin disorders.

Exclusion Criteria:

* Use of systemic or topical antimicrobials during the 2-week pretest conditioning period. This restriction includes but is not limited to shampoos, lotions, soaps, baby powders, and materials, such as solvents, acids, or alkalis.
* A medical diagnosis of a physical condition, which would preclude participation such as: diabetes, hepatitis, an organ transplant, a medical surgical implant, or an immunocompromised system.
* Any medical condition that in the opinion of the investigator would preclude participation.
* Bathed in chemically treated pools or hot tubs 2 weeks prior to any microbial sampling.
* Used UV tanning lamps 2 weeks prior to any microbial sampling.
* Bathing or showering less than 48 hours prior to any microbial sampling.
* Known sensitivity to chlorhexidine gluconate.
* Known sensitivity to latex (rubber).
* Known sensitivity to fragrances.
* Pregnant or nursing.
* Unwillingness to fulfill the performance requirements of the study.
* Subjects who have completed part or all of the study will not be reentered in the study.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 335 (Actual)
Dates: Start 2007-11-13 (Actual); Primary Completion 2008-04-27 (Actual); Study Completion 2008-06-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: M. Hamid Bashir, MD, Principal Investigator — Medical Director
Locations (1):
- Microbiotest, Sterling, Virginia, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Each subject received more than one treatment. Randomization was done by testing site and each subject had 4 testing sites.
Units Other Than Participants: Treated Sites
Groups:
- All Study Participants: Study Participants that were treated
Period: Overall Study
Arm/Group | All Study Participants
Started | 335; 1324 Treated Sites
CHG Swabstick (3 @ Once) | 139; 276 Treated Sites
CHG Swabstick Sequential | 138; 273 Treated Sites
Hibiclens | 133; 264 Treated Sites
Sterile Water Swab (3 @ Once) | 132; 260 Treated Sites
Sterile Water Swabstick (Sequential) | 126; 251 Treated Sites
Completed | 335; 1324 Treated Sites
Not Completed | 0; 0 Treated Sites

BASELINE CHARACTERISTICS:
Population: Participants treated in the study with adequate baseline bacterial load.
Groups:
- All Study Participants: All Participants Who Completed Evaluations
Arm/Group | All Study Participants
Number analyzed (Participants) | 335
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.9 (14.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  All Participants: Female | 149
  All Participants: Male | 186
371-121 Preoperative Skin Preparations [Count of Participants; unit: Participants] — Note: Participants received 2 of the 5 study products. One product is applied to on the left abdomen and groin and one product is applied on the right abdomen and groin.
  Participants
    CHG Swabstick (3 @ Once) | 139
    CHG Swabstick (Sequential) | 138
    Hibiclens | 133
    Sterile Water Swab (3 @ Once) | 132
    Sterile Water Swabstick (Sequential) | 126

OUTCOME MEASURES:

1. Primary Outcome: log10 Reductions From Baseline for Each Test Parameter in CFU (Colony Forming Unit)/cm2 on Inguinal and Abdominal Sites
Description: The bacterial reductions achieved by the test products and the controls using 2 different application techniques at 10-minute and 6-hour sampling intervals for both groin and abdominal sites were evaluated.
Time Frame: 10 minutes and 6 hours after application of test solutions
Population: Measure Analysis Population Description: Number analyzed is not equal to participants treated but rather equal to the number of treated sites for individuals who met the baseline bacterial load criteria on treatment day
Measure: Mean (Standard Deviation); unit: Average log10 reductions in CFU/cm2
Units Other Than Participants: Number of Sites Analyzed
Arm/Group | CHG Swabstick (3 @ Once) | CHG Swabstick Sequential | Hibiclens | Sterile Water Swab (3 @ Once) | Sterile Water Swabstick (Sequential)
Number analyzed (Participants) | 111 | 112 | 111 | 111 | 112
Number analyzed (Number of Sites Analyzed) | 276 | 273 | 264 | 260 | 251
Average log10 reductions in CFU/cm2
  Groin site - 10 minutes: number analyzed (Number of Sites Analyzed) | 111 | 111 | 111 | 111 | 111
  Groin site - 10 minutes | 3.51 (0.62) | 3.44 (0.64) | 3.15 (0.53) | 0.92 (0.47) | 0.97 (0.55)
  Groin site - 6 hours: number analyzed (Number of Sites Analyzed) | 111 | 111 | 111 | 111 | 111
  Groin site - 6 hours | 3.22 (0.65) | 3.24 (0.58) | 2.89 (0.62) | 0.82 (0.47) | 0.85 (0.58)
  Abdomen site - 10 minutes: number analyzed (Number of Sites Analyzed) | 111 | 112 | 111 | 111 | 112
  Abdomen site - 10 minutes | 2.56 (0.50) | 2.58 (0.48) | 2.76 (0.49) | 0.54 (0.37) | 0.50 (0.35)
  Abdomen site - 6 hours: number analyzed (Number of Sites Analyzed) | 111 | 112 | 111 | 111 | 112
  Abdomen site - 6 hours | 2.38 (0.60) | 2.39 (0.64) | 2.51 (0.66) | 0.47 (0.38) | 0.46 (0.39)

ADVERSE EVENTS:
Time Frame: During the study through the 6-hour time point evaluations
Groups:
- CHG Swabstick (3 @ Once): Chlorhexidine gluconate (CHG) 2% CHG/isopropyl alcohol (IPA) 70%-3 swabsticks applied @ same time
  CHG 2% w/v & IPA 70% v/v, swabstick (3 @ once): 3 swabsticks topically applied at the same time to intact skin
- CHG Swabstick Sequential: Chlorhexidine gluconate (CHG) 2% w/v and isopropyl alcohol (IPA) 70% v/v--3 swabsticks applied sequentially
  CHG 2% w/v & IPA 70% v/v swabstick: 3 swabsticks applied sequentially to intact skin.
- Hibiclens: Chlorhexidine gluconate 4% w/v in an aqueous base
  Aqueous CHG 4% w/v applied according to manufacturer's directions: Step 1) 5 mL of Hibiclens applied to a sterile gauze pad. Step 2) Product applied to treatment area on intact skin for 2 minutes. Area dried with sterile towel or sterile gauze. Steps 1 and 2 repeated.
- Sterile Water Swab (3 @ Once): Sterile swabstick wetted with sterile deionized water--3 swabsticks applied at the same time.
  Sterile swabstick with sterile deionized water (3 @ once): 3 swabsticks wetted with sterile water topically applied to intact skin at the same time.
- Sterile Water Swabstick (Sequential): Sterile swabstick wetted with sterile deionized water--3 swabsticks applied sequentially.
  Sterile swabstick with sterile deionized water (sequentially): swabsticks wetted with sterile water topically applied to intact skin sequentially.
Arm/Group | CHG Swabstick (3 @ Once) | CHG Swabstick Sequential | Hibiclens | Sterile Water Swab (3 @ Once) | Sterile Water Swabstick (Sequential)
All-Cause Mortality (participants affected / at risk) | 0/139 | 0/138 | 0/133 | 0/132 | 0/126
Serious Adverse Events (participants affected / at risk) | 0/139 | 0/138 | 0/133 | 0/132 | 0/126
Other Adverse Events (participants affected / at risk) | 0/139 | 0/138 | 0/133 | 0/132 | 0/126

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2007-08-24): https://cdn.clinicaltrials.gov/large-docs/12/NCT00799812/Prot_SAP_000.pdf